CLINICAL TRIAL: NCT03944759
Title: Efficacy of Serratus Anterior Plane Block Using Bupivacaine/Magnesium Sulphate Versus Bupivacaine/Nalbuphine for Mastectomy: a Randomized Double Blinded Comparative Study
Brief Title: Efficacy of Serratus Anterior Plane Block Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: doaa rashwan (Other)
Responsible Party: Sponsor-Investigator, doaa rashwan, Assistant profesor Doaa Rashwan, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMBSURECS/30042019/Ali
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain; Postoperative Complications
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GBM:( bupivacaine/magnesium sulphate) (Active Comparator): serratus plane block will performed in the supine position under strict aseptic conditions before induction of anesthesia.
  GBM:( bupivacaine/magnesium sulphate): will receive bupivacaine 30 ml 0.25 and 500 mg magnesium sulphate
  Interventions: Procedure: serratus anterior plan block
- GBN: ( bupivacaine/nalpuphin) (Active Comparator): serratus plane block will performed in the supine position under strict aseptic conditions before induction of anesthesia.. ( bupivacaine/nalpuphin):received bupivacaine 30 ml 0.25 % and nalpuphine 0.2mg/kg.
  Interventions: Procedure: serratus anterior plan block

INTERVENTIONS:
Procedure: serratus anterior plan block — serratus anterior plan block

SUMMARY:
Breast cancer is the main common cancer among females. . Inadequate control of pain may later develop into chronic pain syndrome (paraesthesias, phantom breast pain, and intercostobrachial neuralgia) in 25-40% of the patients .

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of ultrasound-guided serratus anterior plane block with bupivacaine/ magnesium versus bupivacaine/ nalbuphine in breast cancer surgery.

Patients and methods nclusion criteria:

-ASA I and II female patients, age 25-60 undergoing breast cancer surgery

Exclusion criteria:

* Patient refusal
* Contraindications for regional blocks (eg. Infection at the injection site, coagulopathy)
* Allergy to the drugs used in the study
* Chronic pain therapy,
* BMI more than 30 kg/m2

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II female patients, age 25-60 undergoing breast cancer surgery

Exclusion Criteria:

* -Patient refusal
* Contraindications for regional blocks (eg. Infection at the injection site, coagulopathy)
* Allergy to the drugs used in the study
* Chronic pain therapy,
* BMI more than 30 kg/m2

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
time to first analgesic requirements in minutes | change from base line for 24 hours
  time to first analgesic requirements in minutes by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Rashwan, MD, Study Director — Faculty of Medicine Beni-Suef University
Locations (1):
- Faculty Of Medicine, Beni-Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the protocol
Supporting Information: Study Protocol
Time Frame: after registration for ever
Access Criteria: on the web page
  -